CLINICAL TRIAL: NCT00534937
Title: A Randomized Trial of the Flexitouch Compression System as an Adjunctive Treatment for Venous Stasis Ulcer
Brief Title: Flexitouch Compression System for Venous Stasis Ulcer
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Ineffective Recruitment (Business Decision)
Sponsor: West Penn Allegheny Health System (Other)
Collaborators: The Cleveland Clinic (Other); Tactile Systems Technology, Inc. (Industry)
Responsible Party: Principal Investigator, Satish Muluk, Professor, Surgery, Temple University School of Medicine; Associate Professor, Cardiothoracic Surgery, Drexel University College of Medicine, West Penn Allegheny Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC-4372
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Results first posted 2013-03-01 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-01

CONDITIONS: Venous Stasis Ulcer
Keywords: Venous stasis ulcer; Compression pump; Randomized trial; Flexitouch compression
MeSH Terms: conditions — Varicose Ulcer | interventions — Compression Bandages

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard compression (Active Comparator): Patients in this arm will receive current standard of care (once-weekly short-stretch compression wrapping).
  Interventions: Procedure: Compression wrapping
- Flexitouch (Experimental): Patients in this arm will receive once-a-week short stretch compression wrapping AND once-daily Flexitouch pump application (including Flexitouch application once-a-week in the clinic setting).
  Interventions: Procedure: Flexitouch compression pump

INTERVENTIONS:
Procedure: Compression wrapping — Short-stretch compression wrap will be applied at least once a week.
  Other Names: 3M short-stretch compression wrap
  Arms: Standard compression
Procedure: Flexitouch compression pump — In addition to short-stretch wrapping, this group will received once-daily Flexitouch compression pump, both at home and during the once-a-week clinic visits.
  Other Names: 3M compression wrap
  Arms: Flexitouch

SUMMARY:
The researchers hypothesize that utilization of the Flexitouch system will improve the healing rates of (venous stasis ulcers) VSU compared to traditional compression wrapping therapy alone.

Primary Objective: The primary study objective is to determine whether the complete healing rate of venous stasis ulcers at 12 weeks is improved by the addition of Flexitouch® System compression therapy to a standard regimen of compression wrapping.

Secondary Objectives:

* To determine whether the addition of Flexitouch System compression therapy to a standard regimen of compression wrapping increases the percentage reduction in wound surface area.
* To determine whether the addition of Flexitouch compression therapy to a standard regimen of compression wrapping increases the percentage reduction in volume of the affected limb.
* To determine whether the addition of Flexitouch compression therapy to a standard regimen of compression wrapping decreases the time to healing of the venous stasis ulcer.

DETAILED DESCRIPTION:
Background:

Overview of venous stasis ulcers (1-3): Venous stasis ulceration is a common complication of venous insufficiency in the United States. Venous stasis ulcers (VSU) are associated with very significant morbidity, including patient disability, moderate to severe pain, and frequent leg infections. There is also a large cost associated with the medical care needed for this condition and the inability of patients to work. In some patients, this condition can be life- or limb-threatening.

Current standard of care for VSU: It is widely accepted that VSU should be treated by an individualized program of compression wrapping therapy (3-5). This therapy is designed to counteract the presumed pathophysiology of VSU, which develop as a result of valvular reflux and venous hypertension. However, the efficacy of compression therapy alone is suboptimal, with healing rates of roughly 34% reported after 12 weeks of therapy (6). Various adjunctive treatments have been studied, including artificial skin grafts (6-8). However, none of these adjunctive modalities have become widely accepted for the treatment of VSU.

Potential role of compression pumps: Intermittent sequential compression pumps are widely used as an adjunctive modality in the treatment of VSU. These pumps use high compression and are expensive, but this expense may be outweighed by improved healing of VSU. The use of compression pumps is consistent with the pathophysiology of VSU, but data regarding the efficacy of such therapy is scarce. To date, no study has adequately assessed the efficacy of compression pump therapy in the treatment of VSU (9).

Flexitouch System: The Flexitouch System was designed by a therapist trained in manual lymphatic drainage therapy and is produced by Tactile Systems Technology, Inc. The Flexitouch System was designed to simulate MLD techniques and is intended for home use during the self-management phase of CDT. MLD is one (of four) component(s) of Complete Decongestive Therapy, considered the "Gold Standard" for treatment of lymphedema. MLD is a gentle, manual technique producing very light directional pressure/stretch on the skin with manipulation of healthy lymph nodes and vessels. The effects of properly applied MLD include increased intake of lymphatic loads into the lymphatic system, increased lymphangiomotoricity, increased volume of transported lymph fluid, increased venous return in the superficial venous system, promotion of parasympathetic response and pain control. Treatment is always initiated at the trunk segments, with decongestion of proximal areas, prior to addressing the involved extremity (to clear central areas and promote decongestion of more distal areas). The extremity is then treated in segments, starting with the proximal segments and then progressing from distal to proximal regions. The Flexitouch® System is not intended to replace the intensive phase of CDT. However, it follows the principles of MLD in many ways. Flexitouch system provides limb treatment, but in addition, it addresses trunk congestion. The lower extremity garment set consists of two garments, one garment fits over the affected lower extremity and the other fits over the lower abdomen/trunk. Each garment is made up of multiple inflatable chambers within a flexible, stretchable fabric. The treatment consists of a 2-phase program. As in MLD, the preparation phase begins the treatment starting at the inguinal quadrant. Each curved trunk chamber inflates and deflates sequentially to facilitate the movement of edema fluid into the systemic circulation. The cycle is repeated several times. The inflation/deflation cycle is then repeated in each limb region from the knee to the groin, from the ankle to the knee, and finally from the toes to the ankle. The second phase, drainage, begins the sequential inflation/deflation cycle at the toes and continues moving up the leg to the quadrant of the trunk to facilitate the movement of edema fluid from the inguinal quadrant into the system circulation.

Choice of compression pump device for study of VSU treatment: A variety of inflatable compression pumps are available, but there are no data to help choose among these devices (9). No compression device is accepted as a standard of care for VSU. Flexitouch system differs from standard (intermittent sequential) compression pumps in significant ways. As described above, Flexitouch system is unique as a compression device, because it provides not only sequential limb compression, but also trunk compression. Flexitouch system's two-phase program (preparation and drainage) also makes it different from other compression devices. The fact that the system was created for lymphedema may be an advantage in the treatment of VSU, because many authors (10;11) believe that secondary lymphedema plays an important role among VSU patients.

Study Outline:

Patient enrollment procedure

* An approved consent form and authorization permitting release of personal health information must be signed by the patient or guardian.
* All eligibility requirements indicated in Section 3.0 must be satisfied.
* The patient must be registered by calling the study coordinator Lisa Rudman, at Allegheny General Hospital (412-359-4325).

General treatment plan: After enrollment, all patients will be seen once per week for a 12-week period for standard compression wrapping. At each visit, treatment and assessment will be undertaken as described below. The Flexitouch group only will use the Flexitouch System both at home (once daily) and in-clinic (once per week).

Essential elements of treatment and assessment:

Applicable to ALL patients

* The patients will be seen at the wound center one(1) times per week for 12 weeks.
* Patients will receive compression wrapping as standard of care therapy. The precise amount of compression will be individualized according to patient tolerance using 3M Coban 2 layer Compression System.
* The wound area will be measured and photographed weekly, using wound tracing and planimetry software.
* The limb volume will be measured weekly, using available software (NetHealth, Pittsburgh PA).
* The presence or absence of wound infection will be assessed. The need for wound debridement will be recorded.
* The wound will be scored as to whether or not it has healed. If the wound healed at a previous visit, the presence of recurrent ulceration will be assessed.
* The occurrence of treatment failure will be recorded (see section 7d).
* Comprehensive standard wound care treatment including gentle wound cleansing with saline solution at each visit, maintaining moisture balance in the wound and periwound with appropriate dressings (alginate, foam, hydrogel or hydrocolloid), reminding subjects of the importance of proper nutrition, leg elevation at rest and activity, including frequent ambulation and ankle ROM exercises through the day.

Additional steps applicable to patients randomized to Flexitouch arm:

* Patients will be provided a home Flexitouch unit. They will be given instructions to use the Flexitouch system on a once daily basis. They will not need remove the compression wrap for the home therapy.
* In addition to the home use, at each clinic visit, the patient's trunk and affected limb will be treated for 60 minutes with the Flexitouch system.
* The patient will be asked to indicate their level of comfort with the in-clinic Flexitouch session (scale of 0 to 5; 0 = very comfortable, 5 = very uncomfortable).

ELIGIBILITY:
Inclusion Criteria:

* This study will enroll patients in a prospective manner with chronic venous insufficiency and venous stasis ulceration as determined from clinical presentation, positive venous reflux testing, or both.
* Patients must be 18 years old or more.
* The VSU size must be in the range 1-64 cm2.
* The ulcer must extend through both the epidermis and dermis, with no exposed tendon or bone.
* The VSU must have been present for more than 1 month.
* The ulcer must be located between and including the knee and ankle.
* The wound bed must have viable tissues with granulation tissue.

Exclusion Criteria:

* Exposed bone, tendon, or fascia.
* Severe rheumatoid arthritis.
* History of radiotherapy to the ulcer site.
* Uncontrolled congestive heart failure.
* Receiving corticosteroids or immune suppressives.
* History of collagen vascular disease.
* Known malnutrition (albumin < 2.5 g/dL). If malnutrition is suspected by the principal investigator, the albumin level should be checked to determine whether the patient meets the albumin criterion.
* Ulcer clinically infected at the time of entry into the study. However, patients may be entered into the study after successful treatment of infection.
* Known uncontrolled diabetes (HgbA1c > 12%). If the principal investigator suspects uncontrolled diabetes, the Hgb A1c should be checked to determine patient eligibility.
* Signs of cellulitis, osteomyelitis, or necrotic or avascular ulcer bed(s).
* Known arterial insufficiency (Ankle-brachial index < 0.7, or TCPO2 < 35 mmHg, or Toe brachial index < 0.4). If the principal investigator suspects uncontrolled diabetes, the Ankle-brachial index should be checked to determine patient eligibility.
* Active sickle cell disease.
* Unable to comply with the procedures described in the protocol.
* Enrolled in a clinical evaluation for another investigational wound-care device or drug.
* Patients diagnosed with deep venous thrombosis or phlebitis in the affected limb in the last 6 months.
* Pregnancy, suspected or confirmed.
* History of peripheral vascular disease, or chronic renal disease.
* Known active or recurrent cancer, or currently receiving chemotherapy or radiation therapy.
* History of pulmonary embolism.
* Poorly controlled asthma.
* Use of Apligraf, skin graft or similar biological dressing within 30 days of study entry.
* Patients with concurrent atrophie blanche.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2007-09; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Satish Muluk, MD, Principal Investigator — West Penn Allegheny Health System
Locations (2):
- United States (2):
  - Cleveland Clinic, Cleveland, Ohio
  - Allegheny General Hospital Advanced Wound Healing and Lymphedema Center, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Palfreyman SJ, Nelson EA, Lochiel R, Michaels JA. Dressings for healing venous leg ulcers. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD001103. doi: 10.1002/14651858.CD001103.pub2. PMID 16855958
- [Background] Pascarella L, Schonbein GW, Bergan JJ. Microcirculation and venous ulcers: a review. Ann Vasc Surg. 2005 Nov;19(6):921-7. doi: 10.1007/s10016-005-7661-3. PMID 16247708
- [Background] Black SB. Venous stasis ulcers: a review. Ostomy Wound Manage. 1995 Sep;41(8):20-2, 24-6, 28-30 passim. PMID 7546118
- [Background] Kramer SA. Compression wraps for venous ulcer healing: a review. J Vasc Nurs. 1999 Dec;17(4):89-97; quiz 98-9. doi: 10.1016/s1062-0303(99)90034-1. PMID 10818887
- [Background] Hansson C. Optimal treatment of venous (stasis) ulcers in elderly patients. Drugs Aging. 1994 Nov;5(5):323-34. doi: 10.2165/00002512-199405050-00002. PMID 7833586
- [Background] Mostow EN, Haraway GD, Dalsing M, Hodde JP, King D; OASIS Venus Ulcer Study Group. Effectiveness of an extracellular matrix graft (OASIS Wound Matrix) in the treatment of chronic leg ulcers: a randomized clinical trial. J Vasc Surg. 2005 May;41(5):837-43. doi: 10.1016/j.jvs.2005.01.042. PMID 15886669
- [Background] O'Donnell TF Jr, Lau J. A systematic review of randomized controlled trials of wound dressings for chronic venous ulcer. J Vasc Surg. 2006 Nov;44(5):1118-25. doi: 10.1016/j.jvs.2006.08.004. PMID 17098555
- [Background] Falanga V, Sabolinski M. A bilayered living skin construct (APLIGRAF) accelerates complete closure of hard-to-heal venous ulcers. Wound Repair Regen. 1999 Jul-Aug;7(4):201-7. doi: 10.1046/j.1524-475x.1999.00201.x. PMID 10781211
- [Background] Berliner E, Ozbilgin B, Zarin DA. A systematic review of pneumatic compression for treatment of chronic venous insufficiency and venous ulcers. J Vasc Surg. 2003 Mar;37(3):539-44. doi: 10.1067/mva.2003.103. PMID 12618689
- [Background] Wollina U, Abdel-Naser MB, Mani R. A review of the microcirculation in skin in patients with chronic venous insufficiency: the problem and the evidence available for therapeutic options. Int J Low Extrem Wounds. 2006 Sep;5(3):169-80. doi: 10.1177/1534734606291870. PMID 16928673
- [Background] Felty CL, Rooke TW. Compression therapy for chronic venous insufficiency. Semin Vasc Surg. 2005 Mar;18(1):36-40. doi: 10.1053/j.semvascsurg.2004.12.010. PMID 15791552

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred at medical clinics. The first subject was enrolled in November 2007. The subjects were recruited from current patient populations and new patients coming to the clinic. Advertisement materials were used to increase enrollment with little success.
Groups:
- Flexitouch: Patients in this arm will receive once-a-week short stretch compression wrapping AND once daily Flexitouch pump application (including Flexitouch application once-a-week in the clinic setting).
Period: Overall Study
Arm/Group | Standard Compression | Flexitouch
Started | 42 | 47
Completed | 34 | 35
Not Completed | 8 | 12

BASELINE CHARACTERISTICS:
Groups:
- Standard Compression: Patients in this arm will receive current standard of care (once weekly short-stretch compression wrapping).
- Total: Total of all reporting groups
Arm/Group | Standard Compression | Flexitouch | Total
Number analyzed (Participants) | 42 | 47 | 89
Age Continuous [Mean (Standard Deviation); unit: years] | 56.6 (14.3) | 57.4 (16.1) | 57.0 (15.2)
Sex/Gender, Customized [Number; unit: participants] — The gender of 5 patients was unknown due to incompleted data from a site that was terminated early due to PI relocation.
  participants
    Female | 11 | 12 | 23
    Male | 28 | 33 | 61
    Unknown | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Complete Healing Rate of Venous Stasis Ulcers
Description: Number of subjects that experience complete healing of the study venous stasis ulcer during the 12 week treatment period.
Time Frame: 12 weeks
Measure: Number; unit: participants
Groups:
- Standard Compression: Patients in this arm received current standard of care (once weekly short-stretch compression wrapping).
- Flexitouch: Patients in this arm received once-a-week short stretch compression wrapping AND once-daily Flexitouch pump application (including Flexitouch application once-a-week in the clinic setting).
Arm/Group | Standard Compression | Flexitouch
Number analyzed (Participants) | 42 | 47
participants | 19 | 20

2. Secondary Outcome: Change in Wound Surface Area for Non Healed Subject at 12 Weeks.
Description: Change in wound surface area in cm2 from the initial screening to week 12 for all subject who did not completely healed before or at the 12 week visit.
Time Frame: 12 weeks
Population: The participants are those that didn't achieve complete wound healing after 12 weeks of treatment. The change from screening to week 12 in wound surface area is reported.
Measure: Mean (Standard Deviation); unit: cm2
Groups:
- Flexitouch: Patients in this arm received once-a-week short stretch compression wrapping AND once daily Flexitouch pump application (including Flexitouch application once-a-week in the clinic setting).
Arm/Group | Standard Compression | Flexitouch
Number analyzed (Participants) | 17 | 15
cm2 | -8.1 (9.8) | -9.6 (11.3)

3. Secondary Outcome: Percentage Change in Volume of the Affected Limb (-Reduction; +Increase)
Time Frame: 12 weeks
Population: Number of participants who completed 12 weeks of treatment without healing. Also limb volume measures must have been present.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Standard Compression | Flexitouch
Number analyzed (Participants) | 17 | 16
percentage of change | -2.9 (34.1) | -7 (29.1)

4. Secondary Outcome: Time to Healing of the Venous Stasis Ulcer
Description: Only 2 time points so no calculation details are necessary. The change is calculated as the later time point minus the earlier time point (e.g., 12 weeks minus baseline).
Time Frame: Baseline to 12 weeks
Population: Time to healing can only evaluate the patients that showed healing during the 12 week study therefore the number may not be consistent with other numbers.
Measure: Mean (Standard Deviation); unit: days
Groups:
- Standard Compression: Patients in this arm received current standard of care (once-weekly short-stretch compression wrapping).
Arm/Group | Standard Compression | Flexitouch
Number analyzed (Participants) | 19 | 20
days | 37 (24.9) | 43.9 (22.3)

ADVERSE EVENTS:
Time Frame: AEs were collected form 2007 to 2010 at the time of study closure.
Arm/Group | Standard Compression | Flexitouch
Serious Adverse Events (participants affected / at risk) | 3/42 | 0/47
Other Adverse Events (participants affected / at risk) | 8/42 | 6/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Compression (N=42) | Flexitouch (N=47)
Cellulitis / Infection of lower extremity (Infections and infestations) | 3 (3) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Compression (N=42) | Flexitouch (N=47)
Cellulitis / Infection of lower extremity (Infections and infestations) | 8 (8) | 6 (6)

LIMITATIONS AND CAVEATS:
The study was terminated early due to lack of enrollment which ultimately lead to a limited number of subjects to include in an analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less